CLINICAL TRIAL: NCT01206842
Title: Social Cognition Training in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anja Vaskinn, PhD, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/1538 (REK)
Record Dates: First submitted 2010-09-10; First posted 2010-09-22 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia; Social Cognition
Keywords: functional capacity; training; neurocognition
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- social cognition training (Experimental)
  Interventions: Other: Training in Affect Recognition
- treatment as usual (No Intervention)

INTERVENTIONS:
Other: Training in Affect Recognition — A 12-session social cognitive training programming covering emotion perception and social perception administered in a group setting to up to four participants with schizophrenia at the time
  Arms: social cognition training

SUMMARY:
People with schizophrenia show deficits in social cognition, the ability to process information about other people such as identifying their emotional expressions. Social cognition is associated with everyday life functioning and could therefore be an important treatment target. Several social cognitive training programs have been developed during the last years. Results indicate that social cognitive performance can be ameliorated through commonly used intervention techniques. However, it is less clear whether this improvement generalizes to everyday life. The purpose of this study is to investigate if a social cognitive training program (Training in Affect Recognition) improves performance on social cognitive and neuropsychological tests and leads to improved everyday life functioning in persons with schizophrenia. The study also aims at examining if an improvement is present three months after completion of the training intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 18-55
* diagnosis of schizophrenia or schizoaffective disorder
* IQ > 69
* sufficient mastery of Norwegian to undergo assessments

Exclusion Criteria:

* history of head trauma
* neurological/medical condition known to interfere with central nervous system
* receiving outpatient care at time of recruitment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Social cognitive tests | Within one week and within three months of completed training
  PFA and MASC

SECONDARY OUTCOMES:
Functional capacity tests | Within one week and within three months of completed training
  AIPSS and UPSA-brief
Neuropsychological tests | Within one week and within three months of completed training
  MATRICS

CONTACTS AND LOCATIONS:
Overall Officials: Anja Vaskinn, PhD, Principal Investigator — Oslo University Hospital, Psychosis Research Unit
Locations (1):
- Oslo University Hospital, Oslo, Norway